CLINICAL TRIAL: NCT04403750
Title: Combined Laser-surgical Technology of Rhegmatogenous Retinal Detachment Treatment
Brief Title: Combined Laser-surgical Technology of RRD Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Taevere M.R, Principal Investigator, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Technology of RRD treatment
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined laser-surgical technology (Experimental): Combined laser-surgical technology includes 3 steps:
  1. Nd-YAG laser excision of the vitreoretinal traction zone
  2. Pneumatic retinopexy (10% C3F8)
  3. Barrier laser photocoagulation around retinal break after retinal attachment.
  Interventions: Procedure: Combined laser-surgical technology of RRD treatment

INTERVENTIONS:
Procedure: Combined laser-surgical technology of RRD treatment — 1. Nd-YAG laser excision of the vitreoretinal traction zone
  2. Pneumatic retinopexy (10% C3F8)
  3. barrier laser photocoagulation around retinal break after retinal attachment (2-3 days after pneumatic retinopexy)

SUMMARY:
Purpose: to assess the efficacy and safety of combined laser-surgical technology of RRD treatment

DETAILED DESCRIPTION:
The study takes place in the S.N. Fyodorov "Eye Microsurgery" Federal State Institution located in Moscow, Russian Federation.

The study will include 50 patients with rhegmatogenous retinal detachment due to a horseshoe-tear. In addition to the standard ophthalmological examination, all patients will undergo wide-field optical coherence tomography to determine the extension and localization of the vitreoretinal traction zone. The obtained data will be used to planning the 1st step of laser-surgical treatment. All patients will undergo a combined laser-surgical technology, which includes 3 steps: 1) Nd-YAG laser excision of the vitreoretinal traction zone 2) pneumatic retinopexy (10% C3F8) 3) barrier laser photocoagulation around retinal break after retinal attachment.

The patients are going to be followed up for at least 1 year, the main outcome measures are postoperative primary and final anatomic outcome, BCVA and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Rhegmatogenous retinal detachment extending from the 9-o'clock to the 3-o'clock meridians.
2. Superior retinal break from 9 o'clock to 3 o'clock
3. Single retinal break not greater than 1 clock hours in size
4. Physically and mentally co-operated in post-operative head positioning
5. No (or minimal) proliferative vitreoretinopathy
6. None or mild vitreous hemorrhage.

Exclusion Criteria:

1. Severe concomitant eye pathologies (glaucoma, diabetic retinopathy, macular hole, traumas); OR
2. Ocular media opacities
3. Previous ocular surgeries
4. Age <18 years
5. Previous retinal detachment (index eye)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-06-25 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Retinal reattachment rate | in 1 month after gas resorption
  complete retinal re-attachment

SECONDARY OUTCOMES:
Anatomical success | 3, 6, 12 and 24 months post intervention
  complete retinal re-attachment
Visual acuity | 3, 6, 12 and 24 months post intervention
  ETDRS
Visual acuity | 3, 6, 12 and 24 months post intervention
  Snellen

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Kryl, PhD, MD, Principal Investigator — S.N. Fyodorov Eye Microsurgery State Institution.; Mariiam Taevere, MD, Principal Investigator — S.N. Fyodorov Eye Microsurgery State Institution.; Alexander Doga, Professor, Study Director — S.N. Fyodorov Eye Microsurgery State Institution.
Locations (1):
- The S.N. Fyodorov Eye Microsurgery State Institution., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayzulaeva M.R., Doga A.V., Shkvorchenko D.O., Kryl L.A., Buryakov D.A. [Assessment of peripheral vitreoretinal interface structural changes in patients with local rhematogenous retinal detachments by wide-field optical coherent tomography]. Modern technologies in ophtalmology. 2019 June 25. doi: https://doi.org/10.25276/2312-4911-2019-4-20-23
- [Background] Doga A.V., Shkvorchenko D.O., Kryl L.A., Buryakov D.A., Bayzulaeva M.R. [The assessment of combined laser and microinvasive surgery efficiency in local retinal detachment treatment]. Modern technologies in ophtalmology. 2019 March 20. doi: https://doi.org/10.25276/2312-4911-2019-1-363-368
- See also: Assessment of peripheral vitreoretinal interface structural changes in patients with local rhematogenous retinal detachments by wide-field optical coherent tomography — https://eyepress.ru/article.aspx?40421
- See also: The assessment of combined laser and microinvasive surgery efficiency in local retinal detachment treatment — https://eyepress.ru/article.aspx?30058